CLINICAL TRIAL: NCT03141866
Title: "Determining the Feasibility of Chair-based Physical Activity Interventions, Aimed at Improving Various Aspects of Health and Wellbeing in Geriatric Populations With Pre-existing Frailty, Within a Hospital Ward Setting"
Brief Title: Seated Physical Activity in Ageing
Acronym: SPAA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Birmingham (Other)
Collaborators: The Queen Elizabeth Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: ERN_16-0986S; 675003 (Other Grant/Funding Number: European Commission)
Record Dates: First submitted 2017-04-21; First posted 2017-05-05 (Actual); Last update posted 2019-07-26 (Actual); Status verified 2019-04

CONDITIONS: Frail Elderly Syndrome; Frailty; Physical Activity
MeSH Terms: conditions — Frailty; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Exercise Intervention 1: Move It Or Lose It (MIOLI) (Experimental): An established chair-based physical activity programme for older adults.
  Interventions: Other: Exercise Intervention 1: Move It Or Lose It (MIOLI)
- Exercise Intervention 2: Machine-based resistance training (Experimental): Specialised, chair-based resistance training equipment for older adults.
  Interventions: Other: Exercise Intervention 2: Machine-based resistance training intervention

INTERVENTIONS:
Other: Exercise Intervention 1: Move It Or Lose It (MIOLI) — An established chair-based physical activity programme for older adults.
  Arms: Exercise Intervention 1: Move It Or Lose It (MIOLI)
Other: Exercise Intervention 2: Machine-based resistance training intervention — Specialised, chair-based, pneumatic resistance training equipment for older adults.
  Arms: Exercise Intervention 2: Machine-based resistance training

SUMMARY:
This trial will take the form of a feasibility study; designed to assess the feasibility of a proposed future clinical trial in this setting. This proposed future clinical trial is proposed to assess the impact of physical activity, in the form of specialised chair based physical activity interventions, on the physiological, psychological, cognitive, social and emotional health, and functional capacity of geriatric populations with pre-existing frailty within a clinical hospital ward setting; recognising health as a holistic concept incorporating a multitude of inter-related dimensions. This feasibility study is single-centre (taking place in the Harborne Ward of the Queen Elizabeth Hospital Birmingham, Mindelsohn Way, Edgbaston, Birmingham, United Kingdom).

ELIGIBILITY:
Inclusion Criteria:

* Temporary residents within the Harborne 'living lab' ward of the Queen Elizabeth Hospital Birmingham, Edgbaston, Birmingham, United Kingdom
* ≥ 65 years of age
* Frail according to the Fried Frailty criteria: meeting at least three of the five characteristics of frailty (Fried et al. 2001)
* Have the capacity to speak and read in English
* Anticipated by their care team to remain on the ward for approximately 14 days post enrolment into the study. This will be advised by the patient's care team.

Exclusion Criteria:

* Currently taking part in any other clinical trial which could potentially have an impact upon or influences the findings of the current study
* Currently terminally ill with life expectancy which is less than the duration of the study's interventions
* Severe sensory impairment which would profoundly impact on their capacity to undergo the interventions, even once appropriate adaptations have been made.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2018-09-03 (Actual); Primary Completion 2019-08-09 (Estimated); Study Completion 2019-08-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility | Post-Intervention (2 weeks)
  The primary dependent variable of this feasibility study will relate to the eight primary areas of focus of feasibility studies (Bowen et al. 2009), relating to:
  * Acceptability
  * Demand
  * Implementation
  * Practicality
  * Adaptation
  * Integration
  * Expansion and
  * Limited-efficacy testing
  These eight aforementioned areas (constituting the one variable of feasibility) will serve as the primary dependent variable for this study, in order to establish the feasibility of a proposed future clinical trial within this setting. The dependent variable of feasibility will be assessed through semi-structured interviews with participants post intervention, while focus groups will be utilised with both the intervention implementers and study support staff in order to assess the primary dependent variable of the study. Participant uptake and adherence records will also be employed throughout.

SECONDARY OUTCOMES:
Cortisol (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Dehydroepiandrosterone-sulphate (DHEAS) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Serum cortisol : DHEAS ratio (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
C-reactive proteins (CRP) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Inflammatory Cytokine: Interleukin 6 (IL-6) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Inflammatory Cytokine: Tumor Necrosis Factor alpha (TNFα) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Inflammatory Cytokine: Interferon gamma (IFNy) (Physiological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Hand grip strength (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Leg strength (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Leg power output (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Short Physical Performance Battery (SPPB) (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Katz Index of Independence in Activities of Daily Living (Katz ADL) (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Fried Frailty Phenotype (Functional Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Geriatric Depression Scale (GDS) (Psychological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Hospital Anxiety Depression Scale (HADS) (Psychological Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Standardized Mini-Mental State Examination (SMMSE) (Cognitive Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)
Interpersonal Support Evaluation List (ISEL) (Social Dependent Variable) | Pre-intervention (baseline), and post-intervention (2 weeks)

CONTACTS AND LOCATIONS:
Overall Officials: Prof. Anna Whittaker, Principal Investigator — University of Birmingham
Locations (1):
- Harborne Ward, Queen Elizabeth Hospital Birmingham, Birmingham, West Midlands, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Bowen DJ, Kreuter M, Spring B, Cofta-Woerpel L, Linnan L, Weiner D, Bakken S, Kaplan CP, Squiers L, Fabrizio C, Fernandez M. How we design feasibility studies. Am J Prev Med. 2009 May;36(5):452-7. doi: 10.1016/j.amepre.2009.02.002. PMID 19362699
- [Derived] Doody P, Lord JM, Greig CA, Whittaker AC. Assessing the feasibility and impact of specially adapted exercise interventions, aimed at improving the multi-dimensional health and functional capacity of frail geriatric hospital inpatients: protocol for a feasibility study. BMJ Open. 2019 Nov 21;9(11):e031159. doi: 10.1136/bmjopen-2019-031159. PMID 31753876
- See also: Physical Activity and Nutritional INfluences In ageing (PANINI) project website — http://www.birmingham.ac.uk/generic/panini/index.aspx
- See also: Physical Activity and Nutritional INfluences In ageing (PANINI) project twitter — https://twitter.com/PANINI_EU